CLINICAL TRIAL: NCT05710328
Title: Interim FDG-PET/CT for PreDIcting REsponse of HER2+ Breast Cancer to Neoadjuvant Therapy: DIRECT Trial
Brief Title: Testing the Role of FDG-PET/CT to Predict Response to Therapy Prior to Surgery for HER2-positive Breast Cancer, The DIRECT Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA1211; NCI-2022-10172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA1211 (Other: ECOG-ACRIN Cancer Research Group); EA1211 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; HER2-Positive Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: interventions — Drug Therapy; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (FDG-PET/CT scan) (Experimental): Patients receive FDG IV, undergo PET/CT, receive standard of care chemotherapy, and undergo standard of care surgery on study.
  Interventions: Drug: Chemotherapy; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Chemotherapy — Receive standard of care chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Surgical Procedure — Undergo standard of care surgery
  Other Names: Operation; Surgery; Surgery Type; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial tests how well an imaging procedure called fludeoxyglucose F-18 (FDG) positron emission tomography/computed tomography (PET/CT) works in predicting response to standard of care chemotherapy prior to surgery in patients with HER2-positive stage IIa-IIIc breast cancer. FDG is a radioactive tracer that is given in a vein before PET/CT imaging and helps to identify areas of active cancer. PET and CT are imaging techniques that make detailed, computerized pictures of areas inside the body. The use of FDG-PET/CT may help doctors better decide if a patient needs more or less treatment before surgery in order to get the best response. This study evaluates whether FDG-PET/CT is useful in predicting a patient's response to standard of care chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the negative predictive value (NPV) of neoadjuvant interim (ni)FDG-PET/CT for pathologic complete response (pCR), using delta maximum standardized uptake value corrected for lean body mass day 15 (deltaSULmaxD15), completed through central review, of the primary breast cancer at a threshold of 40%, in patients treated with neoadjuvant HER2-directed therapy.

SECONDARY OBJECTIVES:

I. To estimate the sensitivity, specificity, and positive predictive value (PPV) of niFDG-PET/CT for pCR, using deltaSULmaxD15 of the primary breast cancer at a threshold of 40%, in patients treated with neoadjuvant HER2-directed therapy.

II. To evaluate the performance of niFDG-PET/CT, using deltaSULmaxD15 of the primary breast cancer at a threshold of 40%, as a predictor of 3-year event-free survival (EFS) from time of study registration.

EXPLORATORY OBJECTIVES:

I. To estimate the NPV of niFDG-PET/CT for pCR, using deltaSULmaxD15 of the primary breast cancer at a grid of alternative thresholds ranging from 30% to 60%, in patients treated with neoadjuvant HER2-directed therapy.

II. To compare deltaSULmaxD15 using automated image analysis of FDG-PET/CT by AutoPERCIST (trademark) to standard PET analysis software.

OUTLINE:

Patients receive FDG intravenously (IV), undergo PET/CT, receive standard of care chemotherapy, and undergo standard of care surgery on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients (all genders) must be >= 18 years of age.
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patient must have histologically confirmed HER2-positive primary invasive breast carcinoma by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines that has been determined by local testing.
* Patient must have known (either positive or negative) hormone receptor (estrogen receptor [ER] or progesterone receptor [PR]) status by local testing, per ASCO/CAP guidelines. Patients with either hormone receptor-positive or hormone receptor- negative HER2-positive breast cancer are eligible.
* Patient must have American Joint Committee on Cancer (AJCC) 8th Edition stage IIa-IIIc according to anatomic staging table at diagnosis and below criteria.

  * Patients without nodal involvement (cN0) are eligible if T size > 2.0 cm (T2-4)
  * Patients with nodal involvement (cN1-3) are eligible if T2-4
  * Patients with clinical T4d are not eligible
* Patients with bilateral invasive breast cancers are eligible if both cancers are HER2-positive and at least one meets all protocol eligibility criteria and neither cancer renders the patient ineligible.
* Patients with multiple ipsilateral invasive tumors are eligible as long as all tumors are HER2-positive and at least one tumor focus meets all eligibility criteria. Multiple lesions that appear part of the same index tumor do not require additional biopsy/HER2 testing.
* Patient must plan to start a standard neoadjuvant pertuzumab (or other biosimilars) based regimen.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of this imaging intervention are eligible for this trial.
* Patients with human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* Patient must be participating in the trial at an institution which has agreed to perform the imaging research studies, completed the Eastern Cooperative Oncology Group-American College of Radiology Imaging Network Cancer Center Group (ECOG-ACRIN) defined PET/CT scanner qualification procedures and received ECOG-ACRIN PET/CT scanner approval.

  * For patients who completed the baseline (T0) FDG-PET/CT PRIOR to registration, neoadjuvant pertuzumab-based regimen must start after study registration and within 21 days after the T0 scan.

    * Patients must not have used colony stimulating growth factors within 14 days prior to completing a T0 scan done prior to registration.

Exclusion Criteria:

* Patient must not have any prior treatment for the current breast cancer, including surgery, chemotherapy, hormonal therapy, radiation or experimental therapy.
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the teratogenic effects of FDG in addition to the radiation exposure during PET/CT. All patients of childbearing potential must have a blood test or urine study within 7 days prior to registration to rule out pregnancy.

  * NOTE: A pregnancy test within 7 days prior to the T0 scan is also required but will only need to be done if a) the T0 scan is completed after study registration and b) if the pregnancy test done prior to registration is completed outside of the 7-day window.

A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

* Patient must not have any contraindication to FDG-PET/CT imaging which includes routine glucose values > 200 mg/dL and severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of neoadjuvant interim (ni) fludeoxyglucose F-18 (FDG) positron emission tomography/computed tomography (PET/CT) for pathologic complete response (pCR) | Up to 5 years
  The analysis set for this objective will comprise all patients who enrolled in the study and had a FDG-PET/CT scan at T0 and T1 timepoint. The negative predictive value is defined as the probability that pCR will not be achieved by study participants who experience a using delta maximum standardized uptake value corrected for lean body mass day 15 (deltaSULmaxD15) below 40% and will be estimated via an exact, two-sided 95% confidence interval.

SECONDARY OUTCOMES:
Sensitivity of niFDG-PET/CT for pCR | Up to 5 years
  The analysis set for this objective will be the same as for the primary objective. The estimation approach will also be similar.
Specificity of niFDG-PET/CT for pCR | Up to 5 years
  The analysis set for this objective will be the same as for the primary objective. The estimation approach will also be similar.
Positive predictive value of niFDG-PET/CT for pCR | Up to 5 years
  The analysis set for this objective will be the same as for the primary objective. The estimation approach will also be similar.
Performance of niFDG-PET/CT as predictor of 3-year event-free survival | Up to 5 years
  Using deltaSULmaxD15 of the primary breast cancer at a threshold of 40%. The analysis set for this objective will be the same as for the primary objective. The analysis will compare estimates of 3-year event-free survival between participants with deltaSULmaxD15 above and below the 40% threshold using a log-rank test.

OTHER OUTCOMES:
Negative predictive value of niFDG-PET/CT for pCR | Up to 5 years
  The analytic approach for this objective will parallel the approach for the primary aim for each of selected thresholds in the range from 30% to 60%.
Compare deltaSULmaxD15 using automated image analysis of FDG-PET/CT by AutoPERCIST (trademark) to standard PET analysis software | Up to 5 years
  The analytic approach for this aim will include an assessment of agreement between measures of deltaSULmaxD15 obtained from two methods and an assessment of the negative and positive predictive value of the deltaSULmaxD15 measurement by AutoPERCIST (trademark).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Jacene, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (102):
- United States (97):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - University of Texas at Austin, Austin, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Hennessy MA, Gatsonis C, Jacene H, Connolly RM, Burnette BL, Stringer-Reasor EM, Romanoff J, Taurone A, O'Sullivan CC, Le-Petross HT, Stearns V, Fowler AM, Tang SC, Sepulveda KA, DeMichele AM, Mankoff DA, Wolff AC. EA1211: interim FDG-PET/CT for predicting response of HER2-positive breast cancer to neoadjuvant therapy (DIRECT trial). Future Oncol. 2025 Nov;21(26):3377-3384. doi: 10.1080/14796694.2025.2567840. Epub 2025 Oct 5. PMID 41047708